CLINICAL TRIAL: NCT07197346
Title: The Effects of Repetitive Transcranial Magnetic Stimulation Primed Self-controlled Practice on Motor Learning and Motivation
Brief Title: Repetitive Transcranial Magnetic Stimulation Primed Self-controlled Practice on Motor Learning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, R.O.C. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202506021RINB
Record Dates: First submitted 2025-09-15; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: rTMS Stimulation; Autonomy; Healthy Young Adults
Keywords: motor learning; repetitive transcranial magnetic stimulation; autonomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- iTBS + autonomy (Experimental): Participants receive intermittent theta-burst stimulation (iTBS) as priming, followed by self-controlled practice of a joystick task. The participants will be able to self-select the trials for receiving feedback.
  Interventions: Behavioral: Self-controlled (autonomy); Device: rTMS- iTBS (Intermittent Theta-Burst Stimulation)
- iTBS + Yoked (Active Comparator): Participants receive iTBS priming, then perform motor practice with yoked (non-self-controlled) parameters matched to a self-controlled participant.
  Interventions: Behavioral: Yoked Practice; Device: rTMS- iTBS (Intermittent Theta-Burst Stimulation)
- cTBS + autonomy (Experimental): Participants receive continuous theta-burst stimulation (cTBS) as priming, followed by self-controlled practice of a joystick task. The participants will be able to self-select the trials for receiving feedback.
  Interventions: Device: rTMS - cTBS (Continuous Theta-Burst Stimulation); Behavioral: Self-controlled (autonomy)
- cTBS + Yoked (Active Comparator): Participants receive cTBS priming, then perform motor practice with yoked practice parameters.
  Interventions: Device: rTMS - cTBS (Continuous Theta-Burst Stimulation); Behavioral: Yoked Practice
- Sham + autonomy (Sham Comparator): Participants receive sham TBS stimulation as priming, followed by self-controlled practice of a joystick task. The participants will be able to self-select the trials for receiving feedback.
  Interventions: Behavioral: Self-controlled (autonomy); Device: Sham
- Sham + Yoked (Sham Comparator): Participants receive sham TBS priming, then perform motor practice with yoked parameters.
  Interventions: Device: Sham; Behavioral: Yoked Practice

INTERVENTIONS:
Device: rTMS - cTBS (Continuous Theta-Burst Stimulation) — Continuous theta-burst stimulation (cTBS) is a patterned form of rTMS consisting of bursts of three pulses at 50Hz, repeated every 200ms (5Hz), administered continuously without breaks. In this study, cTBS is delivered over the target cortical area according to established safety guidelines (e.g., a continuous 40s train for a total of 600 pulses) at an intensity set as a percentage of the resting motor threshold. The procedure is used to induce a transient reduction in cortical excitability as a priming intervention prior to motor practice.
  Arms: cTBS + Yoked; cTBS + autonomy
Behavioral: Self-controlled (autonomy) — Self-controlled practice is a motor learning intervention in which participants are granted autonomy to make choices about key aspects of their practice sessions (e.g., when to receive feedback, the sequence/timing of trials, or selection of specific practice parameters). This design allows participants to actively control elements of the training experience according to their preference, thereby fostering intrinsic motivation and engagement. The intervention is grounded in the OPTIMAL theory of motor learning, which highlights the role of autonomy support in enhancing learning outcomes and motivation. In this study, participants in the self-controlled practice group make their own decisions regarding practice conditions, in contrast to yoked controls who follow externally assigned parameters.
  Arms: Sham + autonomy; cTBS + autonomy; iTBS + autonomy
Device: Sham — Sham TBS involves the application of a sham theta-burst stimulation protocol designed to mimic the sensory experience of active TBS without delivering effective magnetic pulses to the brain. This is typically achieved by angling the coil to prevent cortical stimulation. The procedure controls for placebo effects and participant expectations while ensuring blinding. The sham stimulation session matches the timing and setup of active TBS interventions but does not induce cortical excitability changes.
  Arms: Sham + Yoked; Sham + autonomy
Behavioral: Yoked Practice — Yoked practice refers to a motor learning protocol in which participants perform tasks under externally controlled practice conditions, matched to the parameters (e.g., feedback) of a paired participant from a self-controlled practice group. This design removes participant autonomy over practice choices, allowing comparison between self-controlled and externally controlled practice to evaluate the effects of autonomy on motor learning and motivation.
  Arms: Sham + Yoked; cTBS + Yoked; iTBS + Yoked
Device: rTMS- iTBS (Intermittent Theta-Burst Stimulation) — Intermittent theta-burst stimulation (iTBS) is a patterned form of repetitive transcranial magnetic stimulation (rTMS) consisting of bursts of three pulses at 50Hz, repeated every 200ms (5Hz). In this study, iTBS is delivered over the target cortical area using standard protocols (e.g., 2s trains of TBS repeated every 10s for a total of 600 pulses) at an intensity set as a percentage of the resting motor threshold. The procedure aims to facilitate cortical excitability as a priming intervention prior to motor practice.
  Arms: iTBS + Yoked; iTBS + autonomy

SUMMARY:
This study aims to investigate the additive effects of combining self-controlled practice with repetitive transcranial magnetic stimulation (rTMS) pretreatment on motivation enhancement and motor learning performance in healthy young adults. According to the "Optimizing Performance Through Intrinsic Motivation and Attention for Learning" (OPTIMAL) theory, numerous studies have demonstrated that providing learners with autonomy during practice can facilitate intrinsic motivation and motor learning. However, self-controlled practice alone may have limited effects, and further interventions may be required to amplify learning outcomes.

In recent years, non-invasive brain stimulation techniques-particularly high-frequency (facilitatory) rTMS applied to the dorsolateral prefrontal cortex (DLPFC)-have been shown to enhance motivational drive and explicit learning performance by strengthening the connectivity of the DLPFC-midbrain dopamine pathway. For example, 10 Hz high-frequency stimulation can significantly improve learners' accuracy and motivation. Interestingly, several sequence learning studies have found that low-frequency (inhibitory) rTMS, when used as a priming intervention, can instead enhance implicit procedural learning. This effect may occur because inhibiting the lateral prefrontal cortex reduces its top-down suppression of implicit learning systems, thereby releasing procedural learning potential.

Based on the theory of metaplasticity, applying facilitatory or inhibitory stimulation beforehand can alter the threshold of synaptic plasticity, thus influencing subsequent learning outcomes. Therefore, this study designed two DLPFC pretreatments-facilitatory and inhibitory-and combined them with self-controlled practice to systematically examine the interaction between different stimulation protocols on motivation and motor learning.

This cross-sectional experiment plans to recruit 72 healthy participants aged 20 or older, randomly assigned to one of six groups: (1) facilitatory rTMS + self-controlled practice, (2) facilitatory rTMS + yoked control, (3) inhibitory rTMS + self-controlled practice, (4) inhibitory rTMS + yoked control, (5) sham rTMS + self-controlled practice, and (6) sham rTMS + yoked control.

The experiment will last for seven days. On Day 1, participants will complete baseline testing, followed by facilitatory rTMS, inhibitory rTMS, or sham stimulation over the DLPFC. Immediately afterward, they will engage in a trajectory-tracking learning task (manipulating a joystick to reproduce a sine-wave pattern). After practice, participants will complete a motivation assessment. During the trajectory-tracking task, the self-controlled group can choose when to receive feedback to adjust their learning, whereas the yoked control group will receive feedback at time points matched to their paired counterpart.

On Day 2, participants will again receive the assigned rTMS (facilitatory, inhibitory, or sham), complete the trajectory-tracking task, and undergo a motivation assessment. After a five-minute rest, they will perform retention and transfer tests, followed by TMS measurement of cortical excitability. On Day 7, participants will return to the laboratory to complete another retention and transfer test, along with cortical excitability measurement via TMS.

The primary behavioral outcomes are the root mean square error (RMSE) and error estimation (EE) in the trajectory-tracking task. Motivation will be assessed using the Intrinsic Motivation Inventory (IMI). As there have been no prior studies combining DLPFC rTMS pretreatment with practice autonomy, the results of this experimental design are expected to provide new insights and references for enhancing motor learning ability in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18-35 years
2. Right-handed (per Edinburgh Handedness Inventory)
3. Normal or corrected-to-normal vision and hearing
4. Eligible for non-invasive brain stimulation per safety screening (no contraindications to TMS)
5. Able to understand study procedures and provide written informed consent in Chinese
6. Willing to comply with all study visits and tasks, including TBS/rTMS and motor practice
7. For yoked pairing: able to be matched to a counterpart participant for practice parameters

Exclusion Criteria:

1. History of epilepsy, seizures, or unexplained fainting; family history of epilepsy in first-degree relatives
2. Any intracranial metal or implanted medical devices (e.g., cochlear implant, deep brain stimulator, aneurysm clips); non-removable metallic objects in head/neck
3. Cardiac pacemaker or other implanted electronic devices
4. Current or past major neurological or psychiatric disorders (e.g., stroke, traumatic brain injury, multiple sclerosis, major depression, bipolar disorder, schizophrenia)
5. Current use of medications lowering seizure threshold or affecting cortical excitability (e.g., tricyclic antidepressants, bupropion, clozapine, lithium, stimulant or sedative-hypnotic abuse); or unstable psychotropic regimens
6. Active migraine with aura or chronic severe headaches
7. Pregnancy or planning pregnancy during participation; breastfeeding (if your site policy excludes)
8. Substance or alcohol use disorder within the past 12 months; positive alcohol/drug screen on visit days
9. Sleep deprivation (<5 hours) on the day before stimulation, or excessive caffeine (>400 mg) within 6 hours pre-stimulation
10. Dermatologic conditions or open wounds at stimulation or EMG/electrode sites
11. Prior extensive training on the specific motor task used in this study (risk of ceiling effects)
12. Concurrent participation in another interventional study or received brain stimulation (TMS/tDCS) within the past 3 months
13. Any condition that, in the investigator's judgment, makes participation unsafe or data unreliable

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Motor Task Accuracy (Root Mean Square Error, RMSE) | Throughout practice on Day1 and Day2, immediately post-practice on Day2, and at the retention and transfer tests on Day 7.
  Root Mean Square Error (RMSE) on the target motor task, computed across trials within each assessment block to quantify spatial/temporal accuracy. RMSE is calculated as the square root of the mean of squared deviations between the participant's performance trajectory/output and the predefined target/ideal trajectory/output. Lower RMSE indicates better accuracy. The primary endpoint is the change from baseline, defined as RMSE at the post-practice assessment minus RMSE at baseline. If multiple trials are collected per block, RMSE will be averaged across trials to yield a single value per time point. Outliers and artifact-contaminated trials will be handled according to a prespecified quality-control procedure [e.g., exclude trials with >3 SD from block mean or device-detected artifacts], and the number of excluded trials will be recorded.

SECONDARY OUTCOMES:
Intrinsic Motivation Inventory (IMI) | Immediately post-practice on Day 1 and Day 2
  Total IMI score assessing task-related intrinsic motivation (e.g., interest/enjoyment, perceived competence, effort/importance, perceived choice). Specify version, item count, and response scale (e.g., 1-7 Likert). Higher scores indicate higher intrinsic motivation.
Change in Corticospinal Excitability/Inhibition | At baseline before priming, immediately post-practice on Day 2, and on Day 7
  We record Motor Evoked Potential (MEP) Amplitude, Resting and Active Motor Thresholds, Cortical Silent Period (CSP), and Short-Interval Intracortical Inhibition (SICI) via TMS. Resting motor threshold (RMT) and active motor threshold (AMT) determined via standard procedures to anchor stimulation intensities. Peak-to-peak MEP amplitude recorded from the target muscle using single-pulse TMS at fixed intensity relative to resting motor threshold (e.g., 120% RMT). CSP duration measured during tonic contraction using suprathreshold single-pulse TMS. Longer CSP reflects stronger GABA-B-mediated inhibition. Paired-pulse TMS determines SICI with a subthreshold conditioning stimulus followed by a suprathreshold test stimulus at a short interstimulus interval (e.g., 2-3ms). Lower conditioned/test ratio indicates stronger GABA-A-mediated inhibition.
Change in Error Estimation Accuracy (EE) | Post-practice on Day 2, and after tests on Day7
  Subjective estimation of own motor performance error recorded after each trial/block. EE accuracy is defined as the absolute difference between the participant's estimated error and the actual task error (e.g., RMSE) for the same trial/block. Lower values indicate more accurate metacognitive estimation. Outcome is the change from baseline calibration to post-practice.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The IPD collected in this study will be available to other researchers upon reasonable request to the principal investigator after the study has been completed.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The IPD will be available after completion of the study (anticipate to be 2028/12/31) for 7 years (2035/12/31)
Access Criteria: Upon reasonable request to the principal investigator